CLINICAL TRIAL: NCT06216093
Title: Phase I, Randomized, Observer-blind, Placebo-control, Parallel-group, first-in Human Study to Evaluate Safety and Tolerability of EuRSV in Healthy Adults Aged Between 19 Years and 80 Years
Brief Title: Phase I, First-In Human Study to Evaluate Safety and Tolerability of EuRSV in Healthy Adults Aged Between 19 Years and 80 Years
Acronym: EuRSV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EuRSV_101
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Syncytial Virus Infections; Respiratory Syncytial Virus (RSV)
Keywords: EuRSV; RSV; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RSV-1 (Experimental)
  Interventions: Biological: EuRSV
- RSV-2 (Experimental)
  Interventions: Biological: EuRSV
- Normal Saline (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: EuRSV — Healthy adults received 0.5mL single intramuscular dose on Day 0 and Day 28.
  Arms: RSV-1; RSV-2
Other: Placebo Comparator — Healthy adults received 0.5mL single intramuscular dose on Day 0 and Day 28.
  Arms: Normal Saline

SUMMARY:
Phase 1 clinical trial to evaluate the safety of RSV-1 and RSV-2 vaccines in healthy adults aged 19 to 80 years who have voluntarily given written consent to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women who meet the age criteria below
2. Have a body mass index (BMI) of at least 18 Kg/m^2 and no more than 30 Kg/m^2 at the screening visit
3. Women and men of childbearing potential who agree to use a highly effective method of contraception* for the duration of the study (up to 3 months after the last dose of study medication)
4. Agree to refrain from donating blood and transfusions (whole blood, plasma components, platelet components, platelet-plasma components) for the duration of the study.
5. After receiving and understanding a detailed explanation of this clinical trial, voluntarily decide to participate and give written consent.
6. For women of childbearing potential, a negative pregnancy test prior to receiving the investigational drug.

Exclusion Criteria:

1. Clinically significant abnormalities on clinical laboratory tests, electrocardiogram (ECG), or chest x-ray at screening.
2. Positive hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) test results at screening.
3. Have had clinically significant symptoms of respiratory illness within 14 days prior to the first dose of investigational product (e.g., cough, sore throat, dyspnea, wheezing, or nocturnal awakenings due to respiratory symptoms).
4. Active pulmonary infection within 14 days prior to the first dose of investigational medicinal product, or any other significant infectious disease that, in the opinion of the investigator, would render the subject ineligible for participation in the study.
5. Have had an acute febrile illness of 38 celsius degrees or greater within 3 days prior to the first dose of investigational drug
6. Have any of the following conditions, or any serious medical or neuropsychiatric condition that, in the opinion of the investigator, would make them ineligible to participate in this study
7. History of allergic reactions or hypersensitivity to any of the components of the investigational drug.
8. History of serious adverse events, serious allergic reactions, or serious hypersensitivity reactions related to vaccination.
9. History of platelet-related or hemorrhagic disease (such as major venous and/or arterial thrombosis with thrombocytopenia), or history of excessive bleeding or bruising after intramuscular injection or venipuncture, or receiving anticoagulant therapy (except that patients may participate if they are using low-dose anticoagulants (e.g., aspirin <100 mg/day) as determined by the investigator).
10. History of systemic urticaria within 5 years prior to the first dose of investigational drug.
11. Have a history of hereditary or idiopathic angioneurotic edema
12. History of organ or bone marrow transplantation
13. Suspected history of drug abuse or alcohol abuse within 6 months prior to the first dose of investigational medication.
14. History of respiratory syncytial virus (RSV) vaccination or participation in an RSV vaccine clinical trial
15. Treatment with immunosuppressive or immunomodulatory agents or chronic steroid use within 6 months prior to the first dose of investigational product.
16. History of dependent use of antipsychotics or narcotic analgesics within 6 months prior to the first dose of study medication, or psychiatric or social conditions that, in the opinion of the investigator, would make it difficult to comply with the procedures of this study.
17. Received any other investigational drug or received an investigational medical device within 6 months of the screening visit.
18. Treatment with immunoglobulins or blood-derived products within 3 months prior to the first dose of investigational medicinal product or planned treatment during the study period
19. Have received or plan to receive any other vaccine within 4 weeks prior to or after each dose of investigational product.
20. Pregnant or lactating women
21. For any other reason deemed by the investigator to be unsuitable as a patient in this study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events | within 7 days post vaccination
  local and systemic AEs
Occurrence of immediate adverse events | within 30 minutes post vaccination
  local and systemic AEs
Occurrence of unsolicited adverse events | within 52 weeks post vaccination
  local and systemic AEs
Occurrence of serious adverse events | within 52 weeks post vaccination
  local and systemic AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Univsersity Hospital, Seoul, South Korea